CLINICAL TRIAL: NCT04465565
Title: Fluids Administration During Combined Clonidine-Arginine Growth Hormone Stimulation Test- Randomized, 2 Arms, Controlled Study
Brief Title: Fluids Administration During Combined Clonidine-Arginine Growth Hormone Stimulation Test
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RMC068119ctil
Record Dates: First submitted 2020-07-03; First posted 2020-07-10 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2020-06

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone stimulation tests
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, 2 arms, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous fluid administration (Experimental): This arm will include 20 children who received Testoviron or Estrofem prior to the the stimulation test and 40 children who did not receive preparation prior to the stimulation test. Participants in this arm will be treated with I. V of 9%NORMAL SALINE (0. 20cc /Kg) administrated over 60 minutes. The fluids treatment will be initiated 90 minutes after the stimulation test will begin
  Interventions: Procedure: 9% Sodium Chloride (NaCl) IV
- Control Group (No Intervention): This arm will include 20 children who received Testoviron or Estrofem prior to the the stimulation test and 40 children who did not receive preparation prior to the stimulation test. Participants in this arm will not receive fluids intravenously during the stimulation test, unless it will be required due to safety reasons

INTERVENTIONS:
Procedure: 9% Sodium Chloride (NaCl) IV — 9% Sodiun Chloride (NaCl) ( 20cc/kg) adminstrated intravenously
  Arms: Intravenous fluid administration

SUMMARY:
The diagnosis of Growth Hormone deficiency in childhood requires the performance of an artificial pharmacological stimulation tests. There are number of substances that increase the secretion of growth hormone, among them Clonidine and Arginine. One of the possible side effects of both Clonidine and Arginine is a reduction in the blood pressure due to a decreased heart output and declined contraction of peripheral blood vessels. In cases where values of blood pressure at the end of the test are not recovered after two sessions of 15 minutes of physical activity, the patient is treated with I. V of 9%NORMAL SALINE (0. 20cc /Kg) administrated over 30-60 minutes.

The aim of the proposed study is to test whether administration of fluids during the combined Growth Hormone stimulation test Clonidine-Arginine will help in the recovery process from the test (blood pressure > 90/50 mmHg after performing physical activity defined as 15-minutes hike in two consecutive sessions). The study design will be randomized, controlled, 2 arms study.

ELIGIBILITY:
Inclusion Criteria:

* Children referred to combined Arginine- Conidine Growth Hormone stimulation test
* Girls: 7-14 years old and Boys: 7-16 years old
* Weight>20 kg
* Normal thyroid function

Exclusion Criteria:

* BMI over percentile 85
* Genetic syndromes or chromosomal disorders
* Steroid treatment
* Renal failure
* Heart failure

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Average blood pressure | Time 180 mnutes- at time of discharging the participant
  Average blood pressure ( 3 measurements in 5 minutes intervals)

SECONDARY OUTCOMES:
Average blood pressure | Time 0- prior to initiating the Growth Hormone test
  Average blood pressure ( 3 measurements in 5 minutes intervals)
Average blood pressure | Time 90 minutes after completing the Arginine adminstration
  Average blood pressure ( 3 measurements in 5 minutes intervals)
Average blood pressure | Time 150 minutes after completing the Arginine adminstration
  Average blood pressure ( 3 measurements in 5 minutes intervals)
Time elapsed between completing the Growth Hormone test until participant is allowed to go home | Time 180 minutes-at time of discharging the participant (after measuring blood pressure > 50/90mm/Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No